CLINICAL TRIAL: NCT04535609
Title: A Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of 24 Weeks Treatment With REN001 in Patients With Primary Mitochondrial Myopathy
Brief Title: An Efficacy and Safety Study of 24 Week Treatment With Mavodelpar (REN001) in Primary Mitochondrial Myopathy Patients
Acronym: STRIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REN001-201
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Primary Mitochondrial Myopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavodelpar (Experimental): Once daily
  Interventions: Drug: Mavodelpar
- Matched placebo (Placebo Comparator): Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavodelpar — Once daily
  Other Names: REN001
  Arms: Mavodelpar
Drug: Placebo — Once daily
  Arms: Matched placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, multi-centre, study designed to investigate the efficacy and safety of REN001 administered once daily over a 24-week period to patients with PMM.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 years or older with PMM as defined by the International Workshop: Outcome measures and clinical trial readiness in primary mitochondrial myopathies in children and adult (Mancuso et al 2017).
2. A confirmed PMM diagnosis due to known pathogenic gene mutation or deletion of the mitochondrial genome. The Sponsor may authorize local genetic testing at Screening, if required, but results must be available prior to randomization of the subject.
3. Documented PMM primarily characterized by exercise intolerance or active muscle pain.
4. Subjects must be ambulatory and able to perform the walking tests independently (walking aids are allowed).
5. Have no changes to any therapeutic exercise regimen within 30 days prior to Day 1 and be willing to remain on the same therapeutic exercise regimen for the duration of the study.
6. Females should be either of non-child-bearing potential or must agree to use highly effective methods of contraception from Screening through to 30 days after last dose in the study. Males with partners who are WOCBP must also use contraception.
7. Concomitant medications (including supplements) must be stable for at least 1 month prior to enrolment and throughout participation in the study.
8. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion:

1. Participation in a prior REN001 (previously known as HPP-593) study.
2. Currently taking or anticipated to need a PPAR agonist during the study.
3. Subjects with bone deformities or motor abnormalities other than related to the mitochondrial myopathy that may interfere with the outcome measures.
4. Clinically significant kidney disease or impairment calculated as eGFR Grade 2 or above <60ml/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation at Screening.
5. Clinically significant liver disease or impairment of AST or ALT Grade 2 or above (>2.5 x ULN), or Total bilirubin > 1.6 x ULN or >ULN with other signs and symptoms of hepatotoxicity at Screening.
6. Subjects with uncontrolled diabetes and/or a Screening HbA1c of ≥11%.
7. Evidence of significant concomitant clinical disease that may need a change in management during the study or could interfere with the conduct or safety of this study. (Stable well-controlled chronic conditions such hypercholesterolemia, gastroesophageal reflux, or depression under control with medication (other than tricyclic antidepressants), are acceptable provided the symptoms and medications would not be predicted to compromise safety or interfere with the tests and interpretations of this study.)
8. Subjects with a history of cancer. A history of in situ basal cell carcinoma in the skin is allowed.
9. Clinically significant cardiac disease and/or clinically significant ECG abnormalities such as 2nd degree heart block, symptomatic tachyarrhythmia or unstable arrythmia (right bundle branch block, left fascicular block and long PR interval are not excluded) that in the opinion of the Investigator should exclude the subject from completing exercise tests.
10. Evidence of hospitalization for rhabdomyolysis within the year prior to enrolment.
11. Pregnant or nursing females.
12. History of sensitivity to PPAR agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amel Karaa, MD, Principal Investigator — Massachusetts General Hospital (MGH)
Locations (41):
- United States (9):
  - University of California, San Diego, La Jolla, California
  - Myology Institute, University of Florida, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas SouthWestern Medical Center, Dallas, Texas
  - Centre for the Treatment of Pediatric Neurodegenerative Disease, University of Texas McGovern Medical School, Houston, Texas
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - PARC Clinical Research, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - M.A.G.I.C. Clinic (Metabolics and Genetics in Calgary), Calgary, Alberta
  - Adult Metabolic Diseases Clinic, Vancouver General Hospital, Vancouver, British Columbia
- General University Hospital in Prague, Prague, Czechia
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- France (6):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Grand Est
  - Hôpital Roger Salengro, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire d' Angers, Angers, Pays de la Loire Region
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU de Nice, Nice
  - Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region
- Germany (2):
  - University Hospital Bonn Clinic and Polyclinic for Neurology, Bonn
  - Medical Center of the University of Munich Friedrich Baur Institute at the Neurological Clinic and Polyclinic, Munich
- Hungary (2):
  - Semmelweis University Insitute of Genomics and Rare Disorders, Budapest
  - University of Pécs Clinical Centre, Department of Neurology, Pécs
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS Neurophysiopathology Unit, Rome, Lazio
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta" UOC Genetica Medica e Neurogenetica, Milan, Lombardy
  - A.O.U Policlinico di Messina U.O.C Neurologia e Malattie Neuromuscolari, Messina, Sicily
  - Azienda Ospedaliero-Universitaria Pisana Dipartimento di specialita' mediche UOC Neurologia, Pisa, Tuscany
  - IRCCS Istituto delle Scienze Neurologiche, Bologna
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- University of Auckland, Auckland, New Zealand
- Haukeland University Hospital, Bergen, Norway
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (3):
  - Queen Square Centre for Neuromuscular Diseases, London, Greater London
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject completed all screening procedures, was randomized in error and was removed from the study before any study procedures were completed.
Groups:
- Mavodelpar: 100 mg Once Daily
Period: Overall Study
Arm/Group | Mavodelpar | Matched Placebo
Started | 108 | 104
Completed | 100 | 98
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavodelpar | Matched Placebo | Total
Number analyzed (Participants) | 108 | 104 | 212
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 12 | 6 | 18
  26-45 years | 34 | 44 | 78
  46-64 years | 51 | 49 | 100
  =>65 years | 11 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 33 | 28 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 101 | 93 | 194
  Unknown or Not Reported | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  White | 99 | 95 | 194
  Not Reported | 4 | 3 | 7
  Other | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  North America | 17 | 15 | 32
  Australia | 7 | 10 | 17
  Europe | 84 | 79 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change in Distance Walked During a 12 Minute Walk Test
Description: Distance walked in meters
Time Frame: Baseline to Week 24
Population: The full analysis set includes all subjects in the randomized set who received at least one dose of study drug and were not subsequently discontinued from the study for failing eligibility criteria. Subjects were analysed according to the treatment they were assigned at randomization. The FAS was used for baseline analyses and was the primary analysis set for efficacy.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Mavodelpar | Matched Placebo
Number analyzed (Participants) | 106 | 104
meters | 26.75 [12.97 to 40.53] | 30.89 [15.03 to 46.74]

2. Secondary Outcome: Change in PROMIS Short Form - Fatigue 13a (FACIT-fatigue) Scores
Description: The PROMIS is a 13-item questionnaire to describe fatigue and its impact upon daily activities and function. Each item is scored between 1=Not At All and 5=Very Much
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mavodelpar | Matched Placebo
Number analyzed (Participants) | 106 | 104
score on a scale | -0.98 [-2.03 to 0.08] | -2.60 [-3.80 to -1.40]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Regular Investigator assessment
Arm/Group | Mavodelpar | Matched Placebo
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/104
Serious Adverse Events (participants affected / at risk) | 8/108 | 7/104
Other Adverse Events (participants affected / at risk) | 85/108 | 81/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavodelpar (N=108) | Matched Placebo (N=104)
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia Influenza (Infections and infestations) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Nodal Rhythm (Cardiac disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hospitalization (Surgical and medical procedures) | 1 | 0
Cranial Operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavodelpar (N=108) | Matched Placebo (N=104)
COVID-19 (Infections and infestations) | 20 | 13
Diarrhea (Gastrointestinal disorders) | 10 | 3
Nausea (Gastrointestinal disorders) | 10 | 4
Vomiting (Gastrointestinal disorders) | 9 | 5
Refraction Disorder (Eye disorders) | 20 | 15
Fatigue (General disorders) | 7 | 9
Headache (Nervous system disorders) | 10 | 13
Dizziness (Nervous system disorders) | 7 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 11 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Material for public dissemination will be submitted to the Sponsor for review at least 60 days prior to submission for publication, public dissemination, or review by a publication committee. During this period, the Sponsor shall be entitled to make a reasoned request that publication be delayed for a period of up to 6 months from the date of first submission to the Sponsor in order to enable the protection of proprietary information and/or Intellectual Property Rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04535609/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04535609/SAP_001.pdf